CLINICAL TRIAL: NCT06037031
Title: A PHASE 1, OPEN-LABEL, NON-RANDOMIZED, SINGLE-DOSE, PARALLEL GROUP STUDY TO EVALUATE THE PHARMACOKINETICS, SAFETY AND TOLERABILITY OF PF-07923568 IN ADULT PARTICIPANTS WITH RENAL IMPAIRMENT AND HEALTHY ADULT PARTICIPANTS WITH NORMAL RENAL FUNCTION
Brief Title: A Study to Learn How the Body Processes the Study Medicine Called PF-07923568 in People With Loss of Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: C5241016
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — sisunatovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Severe Renal Impairment (Experimental): Participants with severe renal impairment will receive a single oral dose of PF-07923568
  Interventions: Drug: Drug: PF-07923568
- Cohort 2: Normal Renal Function (Experimental): Participants with normal renal function will receive a single oral dose of PF-07923568
  Interventions: Drug: Drug: PF-07923568
- Cohort 3 (Optional): Moderate Renal Impairment (Experimental): Participants with moderate renal impairment will receive a single oral dose of PF-07923568
  Interventions: Drug: Drug: PF-07923568

INTERVENTIONS:
Drug: Drug: PF-07923568 — A single dose of PF-07923568 administered orally as 4 capsules
  Other Names: Sisunatovir

SUMMARY:
The purpose of this study is to understand how the loss of kidney function affects study medicine (PF-07923568) in the body. People with some level of loss of kidney function may process PF-07923568 differently from healthy people. PF-07923568 is developed as a possible treatment for respiratory syncytial virus (RSV) infection. RSV is a common virus that affects the lungs and usually causes mild, cold-like symptoms. RSV can cause severe lung infections in infants, elderly, and adults with other serious medical conditions.

This study is seeking participants who:

* Have less than 25% difference in kidney function between 2 screening visits.
* Meet the eGFR criteria for being assigned to groups. eGFR tells how well the kidney is filtering.
* Are not on hemodialysis. Hemodialysis is a type of treatment that helps the body remove extra fluid and waste products from the blood when the kidneys are not able to.

Participants will take the study medicine as capsules by mouth once at the study clinic. The participants will stay at the study clinic for about 5 days. During that time, the study team will monitor the participants. The study team will take some blood samples to test the level of PF-07923568. This will help us understand if some level of loss of kidney function will have an effect on the study medicine PF-07923568.

ELIGIBILITY:
Inclusion Criteria:

1. Stable renal function defined as ≤25% difference between 2 measurements of absolute estimated glomerular filtration rate (eGFR) during screening.
2. Meet the eGFR criteria for cohort placement during the screening period.
3. Body mass index (BMI) of 16-40 kg/m2; and a total body weight >45 kg (99 lb.).
4. For Cohort 2 Normal Renal Function Group Only: At screening, meet the demographic-matching criteria, including body weight within ±15 kg and age within ±10 years, of the average of the pooled renal impairment cohort.

Exclusion Criteria:

1. Participants with acute renal disease.
2. Participants who are clinically nephrotic.
3. Participants requiring hemodialysis.
4. Renal allograft recipients.
5. Participants who have previously received a kidney, liver, or heart transplant.
6. Urinary incontinence without catheterization.
7. History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HBsAg), or hepatitis C antibody (HCVAb).
8. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
9. Participation in studies of other investigational products (drug or vaccine) at any time during their participation in this study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Baseline through Day 5
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | Baseline through Day 5
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Baseline through Day 5

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline through Day 36
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline through Day 5
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline through Day 5
Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiograms (ECGs) | Baseline through Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Orlando Clinical Research Center, Orlando, Florida
  - Genesis Clinical Research, LLC, Tampa, Florida
  - Prism Research LLC dba Nucleus Network, Saint Paul, Minnesota
  - Clinical Trials of Texas, LLC, San Antonio, Texas
  - Clinical Trials of Texas, LLC dba Flourish Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5241016